CLINICAL TRIAL: NCT02299791
Title: Dissemination of CVD Risk Factor Treatment Among Diabetic Patients in Safety Net Clinics
Acronym: ALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); OCHIN, Inc. (Other); Virginia Garcia Memorial Health Center (Unknown); Multnomah County Health Department (Other Government); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R18HL095481-01A1 (NIH); 1R18HL095481-01A1 (NIH)
Record Dates: First submitted 2014-11-07; First posted 2014-11-24 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases
Keywords: clinic-level interventions; quality improvement; translational medical research; community health centers
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Intervention (Active Comparator): 6 study clinics received the ALL intervention starting 6/1/11
  Interventions: Other: ALL
- Late implementation (Active Comparator): 5 study clinics received the ALL intervention starting 6/1/12
  Interventions: Other: ALL

INTERVENTIONS:
Other: ALL — This clinic-level intervention involves a toolkit of decision support tools. These tools are listed below.
  1. EHR tools to expedite identification
     a. EHR automated point-of-care alerts (Best Practice Alerts)
  2. EHR tools to expedite prescribing
     1. EHR order sets
     2. EHR text shortcuts for notation
     3. patient education materials (handout, poster)
  3. EHR-based outreach support tools a. EHR registries
  Arms: Early Intervention
Other: ALL — These clinics got the same exact intervention, but one year later, as this was a staggered randomized trial.
  Arms: Late implementation

SUMMARY:
The purpose of the ALL Study is to determine the effectiveness of the dissemination of the ALL intervention from an integrated care setting into Community Health Centers (CHCs) by measuring changes in diabetes mellitus (DM) population prescription rates for the medications, using a pre-post comparison within clinics and a staggered, randomized implementation across clinics.

DETAILED DESCRIPTION:
The ALL Initiative ('ALL') is a population-level management program developed at Kaiser Permanente (KP). It seeks to decrease cardiovascular disease (CVD) morbidity and mortality in patients with diabetes by improving rates of prescribing for guideline-concordant cardioprotective medications. Multiple mechanisms supported this intervention at KP. The investigators implemented ALL in 11 Community Health Centers (CHC) in the Portland, Oregon metropolitan area. To our knowledge, this was the first clinical trial testing the translation and implementation of a successful quality improvement (QI) initiative from a private, integrated care setting into CHCs.

The investigators adapted the ALL intervention for CHCs through an iterative, stakeholder-driven process. The investigators then conducted a cluster-randomized pragmatic trial in 11 CHCs in a staggered process with six 'early' CHCs implementing the intervention one year before five 'late' CHCs. The investigators measured monthly rates of cardioprotective prescribing rates. Through segmented regression analysis, the investigators evaluated the intervention's effects in June 2011-May 2013. Participants included 11 CHCs serving ~6,500 adult patients with diabetes mellitus (DM) who were indicated for cardioprotective medications per national guidelines. The investigators also conducted a process evaluation to identify factors important to implementation success.

Our overarching goals were to identify and resolve issues in disseminating a successful program from a large, well-organized health system into CHCs. The investigators hypothesized that cross-setting translation was feasible, and that adapting and implementing proven QI approaches could improve the care CHCs provide without requiring them to develop native initiatives. The investigators anticipated that this implementation would involve substantially adapting potentially 'translatable' practices and interventions, due to the differences between private, integrated care settings and CHCs in terms of patient needs and vulnerability, and system resources.

ELIGIBILITY:
Inclusion Criteria:

* Convenience sample of 11 community health clinics (CHCs) that are members of OCHIN, Inc.

Exclusion Criteria:

* none, for study CHCs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4856 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Gold, PhD, MPH, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gold R, Muench J, Hill C, Turner A, Mital M, Milano C, Shah A, Nelson C, DeVoe JE, Nichols GA. Collaborative development of a randomized study to adapt a diabetes quality improvement initiative for federally qualified health centers. J Health Care Poor Underserved. 2012 Aug;23(3 Suppl):236-46. doi: 10.1353/hpu.2012.0132. PMID 22864500
- [Derived] Gold R, Bunce A, Cowburn S, Davis JV, Hollombe C, Nelson CA, Puro J, Muench J, Hill C, Jaworski V, Mercer M, Howard C, Perrin N, DeVoe J. Cardiovascular care guideline implementation in community health centers in Oregon: a mixed-methods analysis of real-world barriers and challenges. BMC Health Serv Res. 2017 Apr 5;17(1):253. doi: 10.1186/s12913-017-2194-3. PMID 28381249
- [Derived] Gold R, Bunce AE, Cohen DJ, Hollombe C, Nelson CA, Proctor EK, Pope JA, DeVoe JE. Reporting on the Strategies Needed to Implement Proven Interventions: An Example From a "Real-World" Cross-Setting Implementation Study. Mayo Clin Proc. 2016 Aug;91(8):1074-83. doi: 10.1016/j.mayocp.2016.03.014. Epub 2016 Apr 23. PMID 27113199
- [Derived] Gold R, Nelson C, Cowburn S, Bunce A, Hollombe C, Davis J, Muench J, Hill C, Mital M, Puro J, Perrin N, Nichols G, Turner A, Mercer M, Jaworski V, Howard C, Abiles E, Shah A, Dudl J, Chan W, DeVoe J. Feasibility and impact of implementing a private care system's diabetes quality improvement intervention in the safety net: a cluster-randomized trial. Implement Sci. 2015 Jun 10;10:83. doi: 10.1186/s13012-015-0259-4. PMID 26059264
- See also: PubMed — http://www.ncbi.nlm.nih.gov/pubmed?term=Collaborative%20development%20of%20a%20randomized%20study%20to%20adapt%20a%20diabetes%20quality%20improvement%20initiative%20for%20federally%20qualified%20health%20centers%5BTitle%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done at the clinic level. All patients seen in the clinics were potentially eligible for the intervention based on clinic visit and clinical criteria.
Units Other Than Participants: Clinics
Groups:
- Early Intervention Number of Patients: Patients in 6 study clinics received the ALL intervention starting 6/1/11
  ALL: This clinic-level intervention involves a toolkit of decision support tools. These tools are listed below.
  1. EHR tools to expedite identification
     a. EHR automated point-of-care alerts (Best Practice Alerts)
  2. EHR tools to expedite prescribing
     1. EHR order sets
     2. EHR text shortcuts for notation
     3. patient education materials (handout, poster)
  3. EHR-based outreach support tools a. EHR registries
- Late Interventions Number of Patients: 5 study clinics received the ALL intervention starting 6/1/12
  ALL: These clinics got the same exact intervention, but one year later, as this was a staggered randomized trial.
Period: Overall Study
Arm/Group | Early Intervention Number of Patients | Late Interventions Number of Patients
Started | 2053; 6 Clinics | 2803; 5 Clinics
Completed | 2053; 6 Clinics | 2803; 5 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- Early Intervention: 6 study clinics received the ALL intervention starting 6/1/11
  ALL: This clinic-level intervention involves a toolkit of decision support tools. These tools are listed below.
  1. EHR tools to expedite identification
     a. EHR automated point-of-care alerts (Best Practice Alerts)
  2. EHR tools to expedite prescribing
     1. EHR order sets
     2. EHR text shortcuts for notation
     3. patient education materials (handout, poster)
  3. EHR-based outreach support tools a. EHR registries
- Total: Total of all reporting groups
Arm/Group | Early Intervention | Late Implementation | Total
Number analyzed (Participants) | 2053 | 2803 | 4856
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1518 | 2244 | 3762
  >=65 years | 535 | 559 | 1094
Age, Continuous [Mean (Full Range); unit: Years] | 62 [18 to 75] | 63 [18 to 75] | 63 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1240 | 1634 | 2874
  Male | 813 | 1169 | 1982
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 659 | 900 | 1559
  Not Hispanic or Latino | 1374 | 1877 | 3251
  Unknown or Not Reported | 20 | 26 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16 | 22 | 38
  Asian | 101 | 138 | 239
  Native Hawaiian or Other Pacific Islander | 14 | 19 | 33
  Black or African American | 179 | 244 | 423
  White | 1258 | 1717 | 2975
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 485 | 663 | 1148
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2053 | 2803 | 4856

OUTCOME MEASURES:

1. Primary Outcome: Patients Indicated for ACE/ARB and Statin Who Had an Active Prescription for Both
Description: Number of patients indicated for ACE/ARB and statin who had an active prescription for both, as a proportion of patients indicated for ACE/ARB and statin.
Time Frame: Percent of clinic patients prescribed guideline-concordant cardioprotective medications, as of the 1st day of each month, from up to 36 months
Population: clinic patients with diabetes who had a clinic encounter (in person or by telephone) within the previous year and were indicated for ACE/ARB and statin per current national care guidelines
Measure: Count of Participants; unit: Participants
Arm/Group | Early Intervention | Late Implementation
Number analyzed (Participants) | 2053 | 2803
Participants | 1279 | 1318

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored for this cluster randomized trial.
Description: Adverse events were not monitored for this cluster randomized trial.
Arm/Group | Early Intervention | Late Implementation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes